CLINICAL TRIAL: NCT01557400
Title: An Open-Label Study for Previously Treated Ataluren (PTC124®) Patients With Nonsense Mutation Dystrophinopathy
Brief Title: Study of Ataluren for Previously Treated Participants With Nonsense Mutation Duchenne/Becker Muscular Dystrophy (nmDBMD) in Europe, Israel, Australia, and Canada
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-019-DMD
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Dystrophinopathy
Keywords: Duchenne muscular dystrophy; Becker muscular dystrophy; Nonsense mutation; Premature stop codon; DMD; BMD; nmDBMD; DBMD; Ataluren; PTC124
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ataluren (Experimental): Ataluren will be provided as a vanilla-flavored powder to be mixed with water, milk, fruit juice (except apple juice) fruit punch, or in semi-solid food (for example, yogurt, pudding, or applesauce). The dose level for ataluren will be 10 milligrams/kilograms (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening. Administration within 30 minutes after a meal will be recommended. Study drug dosing will be based on milligrams of drug per kilogram of body weight. Because of potential changes in participant body weight over time, weight-based dose adjustment can occur every 24 weeks as required. Study drug will be taken for up to 240 weeks.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Oral powder for suspension
  Other Names: PTC124®

SUMMARY:
Duchenne/Becker muscular dystrophy (DBMD) is a genetic disorder that develops in boys. It is caused by a mutation in the gene for dystrophin, a protein that is important for maintaining normal muscle structure and function. Loss of dystrophin causes muscle fragility that leads to weakness and loss of walking ability during childhood and teenage years. A specific type of mutation, called a nonsense (premature stop codon) mutation, is the cause of DBMD in approximately 10-15% of boys with the disease. Ataluren is an orally delivered, investigational drug that has the potential to overcome the effects of the nonsense mutation. This study comprises a Phase 3, open-label study of ataluren in participants with nmDBMD who previously received ataluren at an Investigator site in a prior PTC-sponsored clinical study. A separate open-label study (PTC124-GD-016-DMD; NCT01247207) is being conducted for nmDBMD participants who previously received ataluren at an Investigator site in the United States (US).

DETAILED DESCRIPTION:
All participating sites must have had at least 1 participant that received ataluren treatment in prior PTC-sponsored clinical studies in DBMD (Phase 2b double-blind, placebo-controlled study [PTC124-GD-007-DMD; NCT00592553] and the subsequent open-label extension study [Study PTC124-GD-007e-DMD; NCT00847379]). It is planned that up to ~96 participants will be enrolled.

It is also planned that participants will receive ataluren 3 times per day (TID) at respective morning, midday, and evening doses of 10 milligrams/kilograms (mg/kg), 10 mg/kg, and 20 mg/kg for approximately 336 weeks. Study assessments will be performed at clinic visits during screening, on the first day of ataluren dosing, and then every 48 weeks during the ataluren treatment period, except for weight, which will be measured every 24 weeks at a primary care physician (PCP).

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of signed and dated informed consent/assent document(s) indicating that the participant (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial. Note: If the study candidate is considered a child under local regulation, a parent or legal guardian must provide written consent prior to initiation of study screening procedures and the study candidate may be required to provide written assent. The rules of the responsible Institutional Review Board/Independent Ethics Committee (IRB/IEC) regarding whether 1 or both parents must provide consent and the appropriate ages for obtaining consent and assent from the participant should be followed.
2. History of exposure to ataluren in a prior PTC study in nmDBMD. Note: Participants are considered eligible only if they received ataluren during their participation in 1 or more prior PTC-sponsored studies of ataluren in nmDBMD. Note: Participants who have participated in a prior or ongoing PTC study with ataluren in nmDBMD at a trial site in the US or Canada, but reside outside of the US and Canada, may be eligible for this study (with the approval of the PTC Therapeutics Medical Monitor).
3. Male sex.
4. In participants who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during ataluren administration and the 6-week follow-up period.
5. Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, laboratory tests, and study restrictions. Note: Psychological, social, familial, or geographical factors that might preclude adequate study participation should be considered.

Exclusion Criteria:

1. Exposure to another investigational drug within 1 month prior to start of study treatment.
2. Eligibility for another ataluren clinical trial that is actively enrolling study participants.
3. Known hypersensitivity to any of the ingredients or excipients of ataluren (Litesse® UltraTM [refined polydextrose], polyethylene glycol 3350, Lutrol® micro F127 [poloxamer 407], mannitol 25C, crospovidone XL10, hydroxyethyl cellulose, vanilla, Cab-O-Sil® M5P [colloidal silica], magnesium stearate).
4. Ongoing use of the following medications:

   1. Coumarin-based anticoagulants (for example, warfarin), phenytoin, tolbutamide, or paclitaxel.
   2. Systemic aminoglycoside therapy
5. Ongoing uncontrolled medical/surgical condition, electrocardiogram (ECG) findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant or make it unlikely that follow-up would be completed.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male participants only are being studied.
Enrollment: 94 (Actual)
Dates: Start 2012-05-20 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — PTC Therapeutics
Locations (21):
- Australia (2):
  - Royal Children's Hospital, Parkville, Melbourne
  - Institute For Neuromuscular Research, The Children's Hospital at Westmead, Westmead
- University Hospital KU Leuven, Leuven, Belgium
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Western Ontario, London, Ontario
- France (3):
  - Hôpital d'Enfants CHU Timone, Marseille
  - Laboratoire d'Exploration Fonctionnelles, Nantes
  - Groupe Hospitalier La Pitie-Salpetriere, Paris
- Germany (2):
  - University of Essen - Clinic for Children, Essen
  - University Hospital, Freiburg im Breisgau
- Hadassah Medical Center, Hebrew University Hospital, Jerusalem, Israel
- Italy (3):
  - Ospedale Maggiore Policlinico in Milan, Milan
  - Ospedale Pediatrico Bambino Gesu, Rome
  - U.O. Complessa di Neuropsichiatria Infantile, Rome
- Spain (2):
  - Hospital Sant Joan de déu, Barcelona
  - Hospital Universitari La Fe, Valencia
- Sweden (2):
  - Queen Silvia Children's Hospital, Gothenburg
  - Astrid Lindgren Pediatric Hospital, Stockholm
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - University of Newcastle Institute of Human Genetics, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Welch EM, Barton ER, Zhuo J, Tomizawa Y, Friesen WJ, Trifillis P, Paushkin S, Patel M, Trotta CR, Hwang S, Wilde RG, Karp G, Takasugi J, Chen G, Jones S, Ren H, Moon YC, Corson D, Turpoff AA, Campbell JA, Conn MM, Khan A, Almstead NG, Hedrick J, Mollin A, Risher N, Weetall M, Yeh S, Branstrom AA, Colacino JM, Babiak J, Ju WD, Hirawat S, Northcutt VJ, Miller LL, Spatrick P, He F, Kawana M, Feng H, Jacobson A, Peltz SW, Sweeney HL. PTC124 targets genetic disorders caused by nonsense mutations. Nature. 2007 May 3;447(7140):87-91. doi: 10.1038/nature05756. Epub 2007 Apr 22. PMID 17450125
- [Background] Hirawat S, Welch EM, Elfring GL, Northcutt VJ, Paushkin S, Hwang S, Leonard EM, Almstead NG, Ju W, Peltz SW, Miller LL. Safety, tolerability, and pharmacokinetics of PTC124, a nonaminoglycoside nonsense mutation suppressor, following single- and multiple-dose administration to healthy male and female adult volunteers. J Clin Pharmacol. 2007 Apr;47(4):430-44. doi: 10.1177/0091270006297140. PMID 17389552
- [Derived] McDonald CM, Muntoni F, Penematsa V, Jiang J, Kristensen A, Bibbiani F, Goodwin E, Gordish-Dressman H, Morgenroth L, Werner C, Li J, Able R, Trifillis P, Tulinius M; Study 019 investigators. Ataluren delays loss of ambulation and respiratory decline in nonsense mutation Duchenne muscular dystrophy patients. J Comp Eff Res. 2022 Feb;11(3):139-155. doi: 10.2217/cer-2021-0196. Epub 2021 Nov 18. PMID 34791888
- See also: 16-2-9 CINRG Listing — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217411&parentIdentifier=PTC124-GD-019-DMD&attachmentIdentifier=0c3d8df5-876e-4f54-9b71-fcb919b589e6&fileName=PTC124-019-CSR-002514_1.0_PTC124-GD-019-DMD_Final_CSR_16-2-9_CINRG_Listing.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The treatment gap between the date of administration of the last dose of ataluren in Study PTC124-GD-007-DMD (NCT00592553) and Study PTC124-GD-007e-DMD (NCT00847379) and the date of administration of the first dose of ataluren in this study (PTC124-GD-019-DMD) ranged from 114.43 to 266.14 weeks (801 to 1863 days).
Pre-assignment Details: Of the 94 enrolled participants, 44 were not ambulatory and 84 were on concomitant therapy with corticosteroids. Participants who were non-ambulatory were not able to run/walk 10 meters in ≤30 seconds at study entry.
Groups:
- Ataluren: Ataluren was provided as a vanilla-flavored powder to be mixed with water, milk, fruit juice (except apple juice) fruit punch, or in semi-solid food (for example, yogurt, pudding, or applesauce). The dose level for ataluren was 10 milligrams/kilograms (mg/kg) in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening. Administration within 30 minutes after a meal was recommended. Study drug dosing was based on milligrams of drug per kilogram of body weight. Because of potential changes in participant body weight over time, weight-based dose adjustment occurred every 24 weeks as required. Study drug was taken for up to 240 weeks.
Period: Overall Study
Arm/Group | Ataluren
Started | 94
Received at Least 1 Dose of Study Drug | 94
Completed | 37
Not Completed | 57
Not completed — Transitioned to Commercial Drug Product | 40
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Ataluren: Ataluren was provided as a vanilla-flavored powder to be mixed with water, milk, fruit juice (except apple juice) fruit punch, or in semi-solid food (for example, yogurt, pudding, or applesauce). The dose level for ataluren was 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening. Administration within 30 minutes after a meal was recommended. Study drug dosing was based on milligrams of drug per kilogram of body weight. Because of potential changes in participant body weight over time, weight-based dose adjustment occurred every 24 weeks as required. Study drug was taken for up to 240 weeks.
Arm/Group | Ataluren
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (2.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 94
Race/Ethnicity, Customized [Number; unit: participants] — Race data were collected, and ethnicity data were not collected in this study.
  participants
    Caucasian | 87
    Asian | 4
    Other | 2
    Unknown/Not Reported | 1
6-Minute Walk Distance (6MWD) as Measured by the 6-Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: meters] — The 6MWD was assessed in participants who were ambulatory using standardized procedures. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test. Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable 6MWT data. Participants who were ambulatory were able to run/walk 10 meters in ≤30 seconds at study entry.
  meters
    number analyzed (Participants) | 49
    (all) | 341.63 (108.106)
Physical Function as Measured by the North Star Ambulatory Assessment (NSAA) [Mean (Standard Deviation); unit: units on a scale] — NSAA: 17 activities, each scored as 0 (activity couldn't be performed), 1 (modified method, achieved goal without assistance), or 2 (normal, achieved goal without assistance). Sum of 17 scores = total score. If fewer than 13 activities were performed, total score was considered missing. If 13-16 activities were performed, total score = sum of scores in x activities that were performed by 17/x. If an activity couldn't be performed due to disease progression/loss of ambulation, a score of 0 was assigned. Linear score was linear transformation of NSAA score to a scale of 0 (worst) to 100 (best). Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable NSAA data. Participants who were ambulatory were able to run/walk 10 meters in ≤30 seconds at study entry.
  units on a scale
    number analyzed (Participants) | 50
    (all) | 19.1 (8.52)
Time to Stand From Supine Position [Mean (Standard Deviation); unit: seconds] — Time to stand from the supine position to a standing position was assessed in ambulatory participants. If the time taken to perform a test exceeded 30 seconds, a value of 30 seconds was used. Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable time to stand from supine data. Participants who were ambulatory were able to run/walk 10 meters in ≤30 seconds at study entry.
  seconds
    number analyzed (Participants) | 38
    (all) | 18.56 (34.349)
Time to Walk/Run 10 Meters [Mean (Standard Deviation); unit: seconds] — Time to walk/run 10 meters was measured in ambulatory participants. If the time taken to perform a test exceeded 30 seconds, a value of 30 seconds was used. Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable data for time to walk/run 10 meters. Participants who were ambulatory were able to run/walk 10 meters in ≤30 seconds at study entry.
  seconds
    number analyzed (Participants) | 50
    (all) | 8.35 (4.693)
Pulmonary Function as Measured by Spirometry [Mean (Standard Deviation); unit: liters] — Pulmonary function parameters of %-predicated forced vital capacity (FVC), percent-predicted forced expiratory volume in 1 second (FEV1), peak expiratory flow (PEF), and peak cough flow (PCF) was assessed in non-ambulatory participants by using a spirometer. Due to the difficulty in obtaining an accurate standing height measurement in non-ambulatory participants, ulna length and arm span were used as a surrogate measure for height when calculating percent-predicted FVC. Population: All enrolled participants who received at least 1 dose of study drug, were non-ambulatory, and had evaluable spirometry data. Participants who were non-ambulatory were not able to run/walk 10 meters in ≤30 seconds at study entry.
  liters
    FVC: number analyzed (Participants) | 39
    FVC | 1.94 (0.509)
    FEV1: number analyzed (Participants) | 35
    FEV1 | 68.60 (18.295)
    PEF: number analyzed (Participants) | 39
    PEF | 9.09 (34.350)
    PCF: number analyzed (Participants) | 25
    PCF | 33.06 (81.985)
Participant and Parent/Caregiver-Reported Activities of Daily Living (ADL), as Measured by EK Scale [Mean (Standard Deviation); unit: units on a scale] — Egen Klassification (EK scale): ordinal scale ranging from 0 (highest level of independent function)-30 (lowest level) points. Scale categories (each scored 0-3): 1) ability to use wheelchair, 2) ability to transfer from wheelchair, 3) ability to stand, 4) ability to balance in the wheelchair, 5) ability to move arms, 6) ability to use hands/arms when eating, 7) ability to turn in bed, 8) ability to cough, 9) ability to speak, and 10) physical well-being. Participant is interviewed to capture how he performs tasks of daily life (Categories 1-9) and how he perceives his wellbeing (Category 10). Population: All enrolled participants who received at least 1 dose of study drug, were non-ambulatory, and had evaluable EK scale data. Participants who were non-ambulatory were not able to run/walk 10 meters in ≤30 seconds at study entry.
  units on a scale
    number analyzed (Participants) | 40
    (all) | 7.8 (3.76)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is any untoward medical occurrence or undesirable event(s) experienced in a participant that begins or worsens following administration of the study drug or study treatment, whether or not considered related to the treatment by the Investigator. A serious adverse event (SAE) was an adverse event (AE) resulting in any of the following outcomes or deemed significant for any other reason, death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), or persistent or significant disability/incapacity not related to nmDBMD. AEs included both SAEs and non-serious AEs. AEs were classified according to National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE) and coded using the Medical Dictionary for Regulatory Activities (MedDRA). A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Week 246
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 94
Participants
  TEAEs | 91
  Treatment-Emergent SAEs | 31
  TEAEs Related to Study Treatment | 26

2. Secondary Outcome: Change From Baseline in 6MWD as Measured by the 6MWT
Description: The 6MWD was assessed in participants who were ambulatory using standardized procedures. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test.
Time Frame: Baseline, Weeks 48, 96, 144, 192, and 240
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable 6MWT data. Participants who were ambulatory were able to run/walk 10 meters in ≤30 seconds at study entry.
Measure: Mean (Standard Deviation); unit: change in meters
Arm/Group | Ataluren
Number analyzed (Participants) | 50
change in meters
  Week 48: number analyzed (Participants) | 42
  Week 48 | -41.71 (48.172)
  Week 96: number analyzed (Participants) | 30
  Week 96 | -76.80 (70.781)
  Week 144: number analyzed (Participants) | 21
  Week 144 | -97.57 (83.761)
  Week 192 | -109.37 (96.238)
  Week 240: number analyzed (Participants) | 8
  Week 240 | -134.16 (94.716)

3. Secondary Outcome: Change From Baseline in Physical Function as Measured by the NSAA
Description: The NSAA was used to evaluate physical function in participants who were ambulatory at study entry, using standardized procedures. The NSAA consisted of 17 activities, each scored as 0 (activity could not be performed), 1 (modified method but achieved goal without physical assistance from another), or 2 (normal, achieved goal without assistance). The sum of these 17 scores was used to form a total score. If fewer than 13 of the 17 activities were performed, the total score was considered missing. If 13 to 16 activities were performed, the total score was calculated by multiplying the sum of the scores in the x activities that were performed by 17/x. If an activity could not be performed due to disease progression/loss of ambulation, a score of 0 was assigned. The linear score was the linear transformation of the NSAA score to a scale of 0 (worst) to 100 (best).
Time Frame: Baseline, Weeks 48, 96, 144, 192, and 240
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable NSAA data. Participants who were ambulatory were able to run/walk 10 meters in ≤30 seconds at study entry.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 50
units on a scale
  Week 48: number analyzed (Participants) | 44
  Week 48 | -2.9 (3.08)
  Week 96: number analyzed (Participants) | 33
  Week 96 | -7.4 (5.61)
  Week 144: number analyzed (Participants) | 23
  Week 144 | -8.8 (6.29)
  Week 240: number analyzed (Participants) | 10
  Week 240 | -13.4 (7.03)

4. Secondary Outcome: Change From Baseline in Time to Stand From Supine Position
Description: Time to stand from the supine position to a standing position was assessed in ambulatory participants. If the time taken to perform a test exceeded 30 seconds or if a participant could not perform the test due to disease progression, a value of 30 seconds was used.
Time Frame: Baseline, Weeks 48, 96, 144, 192, and 240
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable time to stand from supine data. Participants who were ambulatory were able to run/walk 10 meters in ≤30 seconds at study entry.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 50
seconds
  Week 48: number analyzed (Participants) | 30
  Week 48 | 3.33 (5.390)
  Week 96: number analyzed (Participants) | 20
  Week 96 | 6.38 (6.029)
  Week 144: number analyzed (Participants) | 13
  Week 144 | 6.11 (6.798)
  Week 192: number analyzed (Participants) | 10
  Week 192 | 3.84 (8.410)
  Week 240: number analyzed (Participants) | 4
  Week 240 | 11.16 (10.718)

5. Secondary Outcome: Change From Baseline in Time to Walk/Run 10 Meters
Description: Time to walk/run 10 meters was measured in ambulatory participants. If the time taken to perform a test exceeded 30 seconds or if a participant could not perform the test due to disease progression, a value of 30 seconds was used.
Time Frame: Baseline, Weeks 48, 96, 144, 192, and 240
Population: All enrolled participants who received at least 1 dose of study drug, were ambulatory, and had evaluable data for time to walk/run 10 meters. Participants who were ambulatory were able to run/walk 10 meters in ≤30 seconds at study entry.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ataluren
Number analyzed (Participants) | 50
seconds
  Week 48: number analyzed (Participants) | 44
  Week 48 | 1.67 (1.957)
  Week 96: number analyzed (Participants) | 32
  Week 96 | 3.48 (4.481)
  Week 144: number analyzed (Participants) | 23
  Week 144 | 3.07 (2.092)
  Week 192: number analyzed (Participants) | 19
  Week 192 | 3.19 (2.049)
  Week 240: number analyzed (Participants) | 9
  Week 240 | 3.62 (1.858)

6. Secondary Outcome: Change From Baseline in Pulmonary Function as Measured by Spirometry
Description: Pulmonary function parameters of %-predicated FVC, percent-predicted FEV1 (adjusted using ulna length and age), PEF, and PCF was assessed in non-ambulatory participants by using a spirometer. Due to the difficulty in obtaining an accurate standing height measurement in non-ambulatory participants, ulna length and arm span were used as a surrogate measure for height when calculating percent-predicted FVC.
Time Frame: Baseline, Weeks 48, 96, 144, 192, and 240
Population: All enrolled participants who received at least 1 dose of study drug, were non-ambulatory, and had evaluable spirometry data. Participants who were non-ambulatory were not able to run/walk 10 meters in ≤30 seconds at study entry.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Ataluren
Number analyzed (Participants) | 43
liters
  FVC, Week 48: number analyzed (Participants) | 29
  FVC, Week 48 | -0.00 (0.239)
  FVC, Week 96 | -0.06 (0.391)
  FVC, Week 144: number analyzed (Participants) | 25
  FVC, Week 144 | -0.18 (0.422)
  FVC, Week 192: number analyzed (Participants) | 22
  FVC, Week 192 | -0.18 (0.760)
  FVC, Week 240 | -0.24 (0.720)
  FEV1, Week 48: number analyzed (Participants) | 24
  FEV1, Week 48 | -7.98 (10.297)
  FEV1, Week 96 | -11.59 (13.366)
  FEV1, Week 144: number analyzed (Participants) | 20
  FEV1, Week 144 | -20.60 (18.201)
  FEV1, Week 192: number analyzed (Participants) | 21
  FEV1, Week 192 | -19.72 (21.916)
  FEV1, Week 240 | -29.17 (18.759)
  PEF, Week 48: number analyzed (Participants) | 28
  PEF, Week 48 | -7.47 (40.552)
  PEF, Week 96: number analyzed (Participants) | 28
  PEF, Week 96 | 9.67 (78.591)
  PEF, Week 144: number analyzed (Participants) | 25
  PEF, Week 144 | -8.34 (42.763)
  PEF, Week 192: number analyzed (Participants) | 22
  PEF, Week 192 | -9.66 (45.356)
  PEF, Week 240: number analyzed (Participants) | 9
  PEF, Week 240 | -23.77 (70.864)
  PCF, Week 48: number analyzed (Participants) | 22
  PCF, Week 48 | -3.67 (63.604)
  PCF, Week 96: number analyzed (Participants) | 16
  PCF, Week 96 | -14.34 (94.453)
  PCF, Week 144: number analyzed (Participants) | 15
  PCF, Week 144 | -48.51 (102.197)
  PCF, Week 192: number analyzed (Participants) | 14
  PCF, Week 192 | -52.19 (105.178)
  PCF, Week 240: number analyzed (Participants) | 9
  PCF, Week 240 | -81.38 (123.517)

7. Secondary Outcome: Change From Baseline in Participant and Parent/Caregiver-Reported ADL, as Measured by the EK Scale
Description: Activities of daily living after loss of ambulation were measured using the EK scale. The EK scale is an ordinal scale ranging from 0 to 30 points where 0 represents the highest level of independent function and 30 the lowest. The scale consists of 10 categories (each scored 0 to 3), involving different functional domains including 1) ability to use wheelchair, 2) ability to transfer from wheelchair, 3) ability to stand, 4) ability to balance in the wheelchair, 5) ability to move arms, 6) ability to use hands and arms when eating, 7) ability to turn in bed, 8) ability to cough, 9) ability to speak, and 10) physical well-being. The administration of the EK scale consisted of an interview of the participant to capture how he performs the tasks of daily life (as described by Categories 1 to 9) and how he perceives his wellbeing (as described by Category 10). The interviewer observed the participant and assigned the final score for the tasks that could be observed in the clinic.
Time Frame: Baseline, Weeks 48, 96, 144, 192, and 240
Population: All enrolled participants who received at least 1 dose of study drug, were non-ambulatory, and had evaluable EK scale data. Participants who were non-ambulatory were not able to run/walk 10 meters in ≤30 seconds at study entry.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ataluren
Number analyzed (Participants) | 43
units on a scale
  Week 48: number analyzed (Participants) | 35
  Week 48 | 2.0 (3.03)
  Week 96: number analyzed (Participants) | 32
  Week 96 | 2.6 (2.85)
  Week 144: number analyzed (Participants) | 26
  Week 144 | 3.3 (2.31)
  Week 192: number analyzed (Participants) | 26
  Week 192 | 5.3 (2.51)
  Week 240: number analyzed (Participants) | 11
  Week 240 | 7.0 (2.49)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 246
Arm/Group | Ataluren
All-Cause Mortality (participants affected / at risk) | 2/94
Serious Adverse Events (participants affected / at risk) | 31/94
Other Adverse Events (participants affected / at risk) | 88/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=94)
Femur fracture (Injury, poisoning and procedural complications) | 15
Tibia fracture (Injury, poisoning and procedural complications) | 2
Back injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Pneumonia (Infections and infestations) | 3
Actinomycosis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Postoperative abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Ventricular arrhythmia (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=94)
Vomiting (Gastrointestinal disorders) | 28
Abdominal pain upper (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Nasopharyngitis (Infections and infestations) | 40
Gastroenteritis (Infections and infestations) | 19
Upper respiratory tract infection (Infections and infestations) | 19
Influenza (Infections and infestations) | 9
Rhinitis (Infections and infestations) | 9
Lower respiratory tract infection (Infections and infestations) | 8
Ear infection (Infections and infestations) | 7
Respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Disease progression (General disorders) | 27
Pyrexia (General disorders) | 19
Fall (Injury, poisoning and procedural complications) | 21
Femur fracture (Injury, poisoning and procedural complications) | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 7
Joint injury (Injury, poisoning and procedural complications) | 5
Ligament sprain (Injury, poisoning and procedural complications) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Scoliosis (Musculoskeletal and connective tissue disorders) | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 29
Dizziness (Nervous system disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Cardiomyopathy (Cardiac disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 5
Left ventricular dysfunction (Cardiac disorders) | 3
Cardiovascular insufficiency (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 1
Left ventricular hypertrophy (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 4
Influenza like illness (General disorders) | 4
Malaise (General disorders) | 4
Fatigue (General disorders) | 3
Chest pain (General disorders) | 2
Infusion site pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pharyngitis (Infections and infestations) | 4
Fungal infection (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 2
Onychomycosis (Infections and infestations) | 2
Paronychia (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Actinomycosis (Infections and infestations) | 1
Body tinea (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Gastrointestinal viral infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Scarlet fever (Infections and infestations) | 1
Sebaceous gland infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 3
Limb injury (Injury, poisoning and procedural complications) | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 2
Administration related reaction (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Back injury (Injury, poisoning and procedural complications) | 1
Bone fissure (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Chillblains (Injury, poisoning and procedural complications) | 1
Eschar (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1
Spinal cord injury sacral (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Overweight (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Extremity contracture (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Fracture pain (Musculoskeletal and connective tissue disorders) | 2
Muscle contracture (Musculoskeletal and connective tissue disorders) | 2
Spinal deformity (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Lordosis (Musculoskeletal and connective tissue disorders) | 1
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Migraine (Nervous system disorders) | 4
Aphonia (Nervous system disorders) | 1
Hypokinesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 3
Enuresis (Psychiatric disorders) | 3
Sleep disorder (Psychiatric disorders) | 2
Anger (Psychiatric disorders) | 1
Gender dysphoria (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Urine abnormality (Renal and urinary disorders) | 2
Incontinence (Renal and urinary disorders) | 1
Myoglobinuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Strangury (Renal and urinary disorders) | 1
Testicular appendage torsion (Reproductive system and breast disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 3
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Tenotomy (Surgical and medical procedures) | 3
Haemorrhoid operation (Surgical and medical procedures) | 1
Nail operation (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Wedge resection toenail (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Varicose ulceration (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Ear pain (Ear and labyrinth disorders) | 2
Motion sickness (Ear and labyrinth disorders) | 2
Delayed puberty (Endocrine disorders) | 2
Cataract (Eye disorders) | 4
Eye allergy (Eye disorders) | 1
Myopia (Eye disorders) | 1
Cardiac function test abnormal (Investigations) | 3
Cortisol decreased (Investigations) | 3
Weight decreased (Investigations) | 3
Weight increased (Investigations) | 3
Cystatin C increased (Investigations) | 2
Monocyte count decreased (Investigations) | 1
Red blood cells urine (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood corticotrophin decreased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood magnesium increased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Blood testosterone decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Blood urine present (Investigations) | 1
Body temperature increased (Investigations) | 1
Electrocardiogram ST segment elevation (Investigations) | 1
Forced vital capacity decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
High density lipoprotein increased (Investigations) | 1
Lymph node palpable (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Protein urine present (Investigations) | 1
Urinary lipids present (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review.

The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT01557400/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT01557400/SAP_001.pdf